CLINICAL TRIAL: NCT03932045
Title: A Randomized, Subject & Evaluator-blind, Matched Pairs, Prospective Study to Compare the Safety and Efficacy Between SYB Filler (SF-01) and Ellansé M in the Correction of Nasolabial Folds
Brief Title: A Study to Evaluate the Safety and Efficacy of SYB Filler(SF-01) in the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYB-SF01-301
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: A Randomized, Subject & Evaluator-blind, Matched pairs, Prospective Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYB Filler (SF-01) (Experimental): PCL filler
  Interventions: Device: SYB Filler (SF-01)
- Ellansé M (Active Comparator): PCL filler
  Interventions: Device: Ellansé M

INTERVENTIONS:
Device: SYB Filler (SF-01) — Apply up to 1.0 ml of the test device (SF-01) and the contrast device (Ellansé M) to both sides of the nasolabial fold.
  Arms: SYB Filler (SF-01)
Device: Ellansé M — Apply up to 1.0 ml of the test device (SF-01) and the contrast device (Ellansé M) to both sides of the nasolabial fold.
  Arms: Ellansé M

SUMMARY:
The objective of this clinical trial is to verify the safety and efficacy of SYB Filler (SF-01) in the temporary improvement of Nasolabial Folds.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who desire an improvement in the appearance of the nasolabial fold on both sides of the face and who have a score of 3 or 4 on the Wrinkle Severity Rating Scale (WSRS)
2. Individuals who have consented to abstain from any other dermatological procedures or treatments, including treatments for wrinkle reduction in the facial area, during the duration of this study.

Exclusion Criteria:

1. Administered an anticoagulant (with the exception of low dosage aspirin (100mg, up to 300mg/day)) within 2 weeks of the date of the screening
2. Administered Vitamin E or non-steroidal anti-inflammatory drugs or Collagen within 1 week of the date of the screening, or who require these during the period of the study
3. History of bleeding disorder in past or present
4. Received deep-peeling, skin regeneration, plastic surgery (including botulinum toxin injection), wrinkle improvement or acne scar treatment in the facial area within 24 weeks of the date of the screening
5. Administered an hyaluronic acid filler within 24 weeks of the date of the screening

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to 12months in Wrinkle Severity Rating Scale (WSRS) Score by independent evaluator assessed | 12months
  The Wrinkle Severity Rating Scale is a 5-point scale with 1 = Absent; 2 = Mild; 3 = Moderate; 4 = Severe and 5 = Extreme. 1 is the best outcome while 5 is the worst outcome. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon KIM, M.D.,Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea